CLINICAL TRIAL: NCT02429089
Title: Phase I Study of LEE011plus Cetuximab in Patients With Recurrent or Metastatic Squamous Cell Carcinoma of the Head and Neck
Brief Title: Study of LEE011plus Cetuximab in Patients With a Cancer of the Head and Neck
Acronym: CETLEE011
Status: Terminated | Phase: Phase 1 | Type: Interventional
Why Stopped: Decided by the investigator due to the difficulties to recruit
Sponsor: Cliniques universitaires Saint-Luc- Université Catholique de Louvain (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UCL-ONCO 2015-01
Record Dates: First submitted 2015-04-14; First posted 2015-04-29 (Estimated); Last update posted 2020-01-09 (Actual); Status verified 2020-01

CONDITIONS: Squamous Cell Carcinoma of the Head and Neck
Keywords: recurrent; metastatic
MeSH Terms: conditions — Squamous Cell Carcinoma of Head and Neck; Recurrence; Neoplasm Metastasis | interventions — ribociclib

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Group I (Experimental): The patients will receive the same molecules (cetuximab and LEE011) but this phase I study will determine the DLTs by dose escalation of LEE011 (400 mg and 600mg).
  Interventions: Drug: LEE011

INTERVENTIONS:
Drug: LEE011 — The first 12 patients will receive cetuximab associated with LEE011 at doses of 400 mg and 600 mg daily to determine the DLTs and safety.
  In the expansion part, besides safety, objective response rate, progression-free survival and overall survival will be calculated with the inclusion of 14 patients.

SUMMARY:
In this trial, the investigators would like to investigate the activity of LEE011 associated with cetuximab (standard of care for the SCCHN patients at this stade of the disease).

DETAILED DESCRIPTION:
In the mammalian cell cycle, entry into S phase is achieved by cyclin-dependent kinases 4 and 6 (CDK4/6), which activate a family of E2F transcription factors by phosphorylating and deactivating the retinoblastoma protein (pRb). LEE011 is an orally, highly selective small molecule inhibitor of CDK4/6 that potently induces G1 arrest with sub-micromolar IC50's in a variety of pRb-positive cancer cells. A recent study showed that an inhibitor of the CDK4-CCND1 complex showed promising results in SCCHN pre-clinical models. There is a strong rationale to investigate CDK inhibitors in this disease. In phase Ib/II study as a single agent, the major toxicities observed were Grade 3 and 4 fatigue (53.8%), nausea (50.8%), neutropenia (47.7%), anemia (37.1%), leukopenia (46.2%), thrombocytopenia (34.1%), diarrhea (32.6%), vomiting (34.8%), lymphocytes count decreased (30.3%), anorexia (21.2%), hyperglycemia (21.2%), constipation (19.7%), hypoalbuminemia (18.9%), dyspnea (18.2%) and cough (16.7%).

ELIGIBILITY:
Inclusion Criteria:

1. Recurrent and/or metastatic head and neck squamous cell carcinoma not amenable to curative treatment with surgery and/or chemotherapy and/or radiation.
2. HPV negative tumors
3. Previous treatment with anti-EGFR based therapy is allowed
4. Measurable disease, i.e., at least one measurable lesion as per RECIST 1.1 criteria (Tumor lesions previously irradiated or subjected to other locoregional therapy will only be considered measurable if disease progression at the treated site after completion of therapy is clearly documented).
5. Progressive disease within 1 year after first line platinum-based chemotherapy given either as a part of the multimodal curative treatment or in the palliative setting or patients non-eligible for platinum therapy.
6. Tumor easily accessible for a biopsy
7. ECOG performance status 0-1, in stable medical condition
8. Patients must have an expected survival of at least 3 months.
9. Paraffin-embedded tumor tissue available for immunohistochemistry
10. Patients must be over 18 years old and must be able to give written informed consent.
11. Women of child-bearing age or sexually active female patients with reproductive potential must have a negative pregnancy test (serum or urine within the 7 days prior to enrollment).
12. Patients able to swallow ribociclib capsules / tablets
13. Patient has adequate bone marrow and organ function as defined by the following laboratory values :

    1. Absolute neutrophil count ≥ 1.5 × 109/L.
    2. Platelets ≥ 100 × 109/L.
    3. Hemoglobin ≥ 9 g/dl.
    4. Potassium, total calcium (corrected for serum albumin), magnesium, sodium and phosphorus within normal limits for the institution or corrected to within limits with supplements before first dose of study medication.
    5. INR ≤ 1.5.
    6. Serum creatinine ≤ 1.5 × mg/dL or creatinine clearance ≥50 mL/min.
    7. In the absence of liver metastases, Alanine aminotransferase (AST) and aspartate aminotransferase (ALT) ≤ 2.5x ULN. If the patient has liver metastases, ALT and AST < 5 x ULN.
    8. Total serum bilirubin ≤ ULN; or total bilirubin ≤ 3.0 x ULN or direct bilirubin ≤1.5 x ULN in patients with well documented Gilbert's Syndrome.
14. Signed informed consent prior to beginning protocol specific procedure.

Exclusion Criteria:

1. Non-squamous head and neck cancer
2. Nasopharynx cancer
3. Patient who received any CDK4/6 inhibitor.
4. Patient has a known hypersensitivity to any of the excipients of LEE011 (ribociclib) or combination drug
5. Patient is concurrently using other anti-cancer therapy.
6. Patient has had major surgery within 14 days prior to starting study drug or has not recovered from major side effects (tumor biopsy is not considered as major surgery).
7. Patient who has not had resolution of all acute toxic effects of prior anti-cancer therapy to NCI CTCAE version 4.03 Grade <1 (exception to this criterion: patients with any grade of alopecia are allowed to enter the study).
8. Patient who has received radiotherapy ≤ 4 weeks or limited field radiation for palliation ≤ 2 weeks prior to starting study drug, and who has not recovered to grade 1 or better from related side effects of such therapy (with the exception of alopecia) and/or from whom ≥ 25% (R. E. Ellis 1961) of the bone marrow was irradiated.
9. Patient has a concurrent malignancy or malignancy within 3 years prior to starting study drug, with the exception of adequately treated, basal or squamous cell carcinoma, non-melanomatous skin cancer or curatively resected cervical cancer.
10. Patients with central nervous system (CNS) involvement unless they meet ALL of the following criteria:

    * At least 4 weeks from prior therapy completion (including radiation and/or surgery) to starting the study treatment
    * Clinically stable CNS tumor at the time of screening and not receiving steroids and/or enzyme-inducing anti-epileptic medications for brain metastases.
11. Patient has impairment of gastrointestinal (GI) function or GI disease that may significantly alter the absorption of the study drugs (e.g., ulcerative diseases, uncontrolled nausea, vomiting, diarrhea, malabsorption syndrome, or small bowel resection)
12. Patient has a known history of HIV infection (testing not mandatory)
13. Patient has any other concurrent severe and/or uncontrolled medical condition that would, in the investigator's judgment, cause unacceptable safety risks, contraindicate patient participation in the clinical study or compromise compliance with the protocol (e.g. chronic pancreatitis, chronic active hepatitis, active untreated or uncontrolled fungal, bacterial or viral infections etc.)
14. Patient has active cardiac disease or a history of cardiac dysfunction including any of the following:

    * History of acute coronary syndromes (including myocardial infarction, unstable angina, coronary artery bypass grafting, coronary angioplasty or stenting) or symptomatic pericarditis within 12 months prior to screening.
    * History of documented congestive heart failure (New York Heart Association functional classification III-IV)
    * Documented cardiomyopathy
    * Patient has a Left Ventricular Ejection Fraction (LVEF) < 50% as determined by Multiple Gated acquisition (MUGA) scan or echocardiogram (ECHO)
    * History of any cardiac arrhythmias, e.g., ventricular, supraventricular, nodal arrhythmias, or conduction abnormality in the previous 12 months of screening.
    * On screening, any of the following cardiac parameters: bradycardia (heart rate < 50 at rest), tachycardia (heart rate > 90 at rest), PR interval > 220 msec, QRS interval >109 msec, or QTcF >450 msec.
    * Congenital long QT syndrome or family history of long QT syndrome
    * Systolic blood pressure >160 or <90 mmHg at screening
    * Bradycardia (heart < 50 at rest), by ECG or pulse, at screening
15. On screening, inability to determine the QTcF interval on the ECG (i.e.: unreadable or not interpretable) or QTcF >450 msec (using Fridericia's correction). All as determined by screening ECG (mean of triplicate ECGs)
16. Patient with a Child-Pugh score B or C
17. Patient is currently receiving any of the following medications and cannot be discontinued 7 days prior to the start of the treatment (see Appendix 1 for details):

    * That are known strong inducers or inhibitors of CYP3A4/5. including grapefruit, grapefruit hybrids, pummelos, star-fruit, and Seville oranges
    * That have a known risk to prolong the QT interval or induce Torsades de Pointes.
    * That have a narrow therapeutic window and are predominantly metabolized through CYP3A4/5.
    * Herbal preparations/medications, dietary supplements
18. Patient is currently receiving or has received systemic corticosteroids ≤ 2 weeks prior to starting study drug, or who have not fully recovered from side effects of such treatment.

    • The following uses of corticosteroids are permitted: single doses, topical applications (e.g., for rash), inhaled sprays (e.g., for obstructive airways diseases), eye drops or local injections (e.g., intra-articular)
19. Patient is currently receiving warfarin or other coumarin-derived anticoagulant for treatment, prophylaxis or otherwise. Therapy with heparin, low molecular weight heparin (LMWH) or fondaparinux is allowed.
20. Participation in a prior investigational study within 30 days prior to enrollment or within 5 half-lives of the investigational product, whichever is longer
21. Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception throughout the study and for 8 weeks after study drug discontinuation. Highly effective contraception methods include:

    * Total abstinence when this is in line with the preferred and usual lifestyle of the patient. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception
    * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
    * Male sterilization (at least 6 months prior to screening). For female patients on the study, the vasectomized male partner should be the sole partner for that patient
    * Combination of any of the two following (a+b or a+c or b+c)

      1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception
      2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
      3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/ vaginal suppository In case of use of oral contraception, women should have been stable on the same pill before taking study treatment.

    Note: Oral contraceptives are allowed but should be used in conjunction with a barrier method of contraception due to unknown effect of drug-drug interaction.

    Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.]
22. Sexually active males unless they use a condom during intercourse while taking the drug and for 30 days after stopping treatment and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.
23. Patient has a history of non-compliance to medical regimen or inability to grant consent.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Actual)
Dates: Start 2015-04; Primary Completion 2017-09-01 (Actual); Study Completion 2018-09-01 (Actual)

PRIMARY OUTCOMES:
To determine the maximum tolerated dose | Up to 20 months

SECONDARY OUTCOMES:
To evaluate the toxicity profile (with CTCAE 4.03 scale) | Up to 20 months

CONTACTS AND LOCATIONS:
Overall Officials: Institut Roi Albert II Cliniques universitaires Saint-Luc, Study Director — Institut Roi Albert II, Cliniques universitaires Saint-Luc
Locations (5):
- Belgium (5):
  - Grand Hôpital de Charleroi site Notre Dame, Charleroi, Hainaut
  - Hôpital de Jolimont, Haine-Saint-Paul, Hainaut
  - Cliniques universitaires Saint-Luc, Brussels
  - Universitair Ziekenhuis Gent, Ghent
  - Clinique et Maternité Sainte-Elisabeth, Namur

REFERENCES:
- [Derived] Seront E, Schmitz S, Papier M, van Maanen A, Henry S, Lonchay C, Rottey S, van Caloen G, Machiels JP. Phase 1 Study Evaluating the Association of the Cyclin-Dependent Kinase 4/6 Inhibitor Ribociclib and Cetuximab in Recurrent/Metastatic p16-Negative Squamous Cell Carcinoma of the Head and Neck. Front Oncol. 2019 Mar 19;9:155. doi: 10.3389/fonc.2019.00155. eCollection 2019. PMID 30941307